CLINICAL TRIAL: NCT00411944
Title: Prospective Study of the Influence of CYP3A4/CYP3A5 and MDR1 Gene Single Nucleotide Polymorphisms on Long-Term Tacrolimus Disposition in Renal Allograft Recipients: a Five Year Follow-up Study Using Abbreviated Concentration-Time Measurements.
Brief Title: Long-Term Pharmacokinetics of Tacrolimus in Renal Recipients
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Other Study IDs: TacLTPK
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-12

CONDITIONS: Renal Transplantation
Keywords: tacrolimus pharmacokinetics; CYP3A4 - CYP3A5; P-glycoprotein; single nucleotide polymorphisms; renal transplantation; calcineurin-inhibitor-associated nephrotoxicity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
An evaluation of the effects of genetically determined variant metabolizing and transporting proteins involved in the disposition of the immunosuppressive drug tacrolimus in renal transplant recipients. In a five year follow-up study tacrolimus dose-corrected exposure changes significantly and the effect(s) of single nucleotide polymorphisms of the CYP3A4/CYP3A5 and MDR1 genes on the latter is assessed in this study.

DETAILED DESCRIPTION:
A 5-year pharmacokinetic follow-up study in 95 renal allograft recipients assessing tacrolimus exposure using repeated abbreviated Area-Under-the-Concentration-time (AUC) curve measurements at regular time points after grafting. The effects of the CYP3A5*1, CYP3A4*1B, MDR1 G2677T/A and C3435T single nucleotide polymorphisms on the evolution of tacrolimus disposition are studied over 5 years in order to clarify the interrelationship between CYP3A5, CYP3A4 and MDR1 genotypes, time-dependent exposure and tacrolimus-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary single kidney transplantation
* Age older than 18 yrs

Exclusion Criteria:

* Combined organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1999-08; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Dirk R Kuypers, MD, PhD, Principal Investigator — Dpt Nephrology and Renal Transplantation, University Hospitals Leuven, Belgium
Locations (1):
- Department of Nephology and Renal Transplantation, Leuven, Belgium

REFERENCES:
- [Result] Kuypers DR, Claes K, Evenepoel P, Maes B, Coosemans W, Pirenne J, Vanrenterghem Y. Time-related clinical determinants of long-term tacrolimus pharmacokinetics in combination therapy with mycophenolic acid and corticosteroids: a prospective study in one hundred de novo renal transplant recipients. Clin Pharmacokinet. 2004;43(11):741-62. doi: 10.2165/00003088-200443110-00005. PMID 15301578
- [Result] Kuypers DR, Claes K, Evenepoel P, Maes B, Vanrenterghem Y. Clinical efficacy and toxicity profile of tacrolimus and mycophenolic acid in relation to combined long-term pharmacokinetics in de novo renal allograft recipients. Clin Pharmacol Ther. 2004 May;75(5):434-47. doi: 10.1016/j.clpt.2003.12.009. PMID 15116056